CLINICAL TRIAL: NCT03358316
Title: Correlation Analysis Between Rotator Cuff Tear and the Superior Migration of Humeral Head
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Yichong, Department of orthopaedics and trauma, Peking University People's Hospital
Other Study IDs: PKUPH-CRT
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear; Magnetic Resonance Imaging; humeral migration
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cuff tear patients: Patients with cuff tear

SUMMARY:
To evaluate the association between rotator cuff tear and the proximal migration of humeral head

DETAILED DESCRIPTION:
In this research, 60 patients with unilateral rotator cuff tear in Peking University People's Hospital in 2018 are planned to be recruited .They will receive Magnetic Resonance Imaging(MRI) and X-ray of the painful shoulder before enrollment in this study, the duration between the two examinations was no longer than 1 week, also there is no past history of surgery in the selected shoulders. There is no other exclusion criteria. Upward Migration Index(UMI) is the ratio between the distance of humeral head center to the lower surface of acromion, and the radius of humeral head circle. It can help to minimize the effect of anatomy difference and imaging magnification, compared with the traditional acromiohumeral distance(AHD). Then we use the Spearman correlation analysis to evaluate the relationship between UMI and fatty degeneration, rotator cuff tear size and the thickness of ruptured supraspinatus tendon from X-ray and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient receive Magnetic Resonance Imaging half year before enrollment, showing supraspinatus tear
* Patient receive X-ray half year before enrollment
* the duration between the two examinations was no longer than 1 week
* no past history of surgery in the selected shoulders

Exclusion criteria:

* patients who cannot receive MRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 60 patients with cuff tear
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between rotator cuff tear size and the superior migration of humeral head | 1 year
  Correlation between rotator cuff tear size and the superior migration of humeral head

SECONDARY OUTCOMES:
Correlation between rotator cuff fatty degeneration and the superior migration | 1 year
  Correlation between rotator cuff fatty degeneration and the superior migration

CONTACTS AND LOCATIONS:
Overall Officials: Yichong Zhang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No